CLINICAL TRIAL: NCT04989270
Title: A Five-year Retrospective Study to Find a Superior Anesthetic Technique for the Cesarean Section From a Hemodynamic Perspective.
Brief Title: A Superior Anesthetic Technique for the Cesarean Section From a Hemodynamic Perspective.
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Other Study IDs: MREC#2178
Record Dates: First submitted 2021-07-05; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-05

CONDITIONS: Obstetric Anaesthesia With Cardiac Complications
Keywords: cesarean section; hemodynamics; general anesthesia; regional anesthesia; intraoperative complications; APGAR Score
MeSH Terms: conditions — Intraoperative Complications | interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Cesarean section: Group of patients undergoing Cesarean section between Jan'2015 to Dec'2019
  Interventions: Procedure: General Anesthesia; Procedure: Regional Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — General anesthesia with intubation, ventilation, intravenous and inhalational anesthetics, opioids and muscle paralysis
Procedure: Regional Anesthesia — Spinal Anesthesia, Epidural Anesthesia

SUMMARY:
Cesarean section operations are increasing in rates worldwide. A proper anesthetic technique is required to maintain the safety of both the mother and the fetus. This study examines the adverse hemodynamic effects associated with general and regional anesthesia and proposes a superior technique from the hemodynamic perspective.

A retrospective cohort study with a five-year study period was conducted on patients who underwent cesarean section with general anesthesia (GA) and regional anesthesia (RA) after obtaining ethical committee approval. Data (hypotension, bradycardia, and blood loss) was collected from hospital information system records of the patients who underwent cesarean section from January 2015 to December 2019. The significance of the variables was determined using the Chi-square test.

A total of 2500 patients were studied. 1379 patients underwent cesarean section with RA meanwhile 1121 patients with GA.

DETAILED DESCRIPTION:
Cesarean section Over the past few decades, cesarean section (CS) rates have been increasing tremendously; it is the most called for surgery in the obstetric department, for instance; in the US, there was an increase of CS by 14% from 1998 to 2001 with a 53% increase in elective primary CS rates and a 13% increase in medically advised primary CS rates (Alnour et al., 2015). The term primary CS is used when the operation is done for the first time on a pregnant patient (Saha and Chowdhury, 2011). This increase in CS rates can be explained by the increased demand for the comfort aspect during labor and the lifesaving properties of this operation in certain conditions for both the mother and the baby (Chen et al., 2019; Tadevosyan et al., 2019). A superior anesthetic method should ease surgical discomfort, decrease postoperative adverse effects, and should have excellent intraoperative analgesia (Alnour et al., 2015; Chen et al., 2019). An anesthetic is used to alleviate the pain of CS operation using either general (GA) or regional (RA) (spinal (SA) and epidural (EA)) anesthetics; sometimes, they can be used together (Alnour et al., 2015).

Pregnancy-induced hypotension The physiological changes associated with pregnancy and aortocaval compression or supine hypotension syndrome are the primary cause of hypotension during pregnancy (Mavridou et al., 2013). Aortocaval compression associated with natural pregnancy decreases cardiac output (CO) and venous return (VR). It starts at 20 weeks of gestation when the patient is lying flat in the supine position. Blood flow from the lower extremities will be disrupted and delayed from reaching the central circulation and the maternal heart; this happens due to the compression force applied by the uterus on the inferior vena cava and the abdominal aorta. This could restrain blood flow to the uterus, increases the risk of morbidity and mortality for both the mother and the fetus. Therefore, choosing a proper anesthetic technique that will not cause further hypotension during the process of CS is important (Mavridou et al., 2013; Alnour et al., 2015; Šklebar et al., 2019).

Anesthesia-induced hypotension There are two definitions of anesthesia-induced hypotension based on studies. It is a decrease to 80% from the baseline blood pressure value or a decrease of systolic arterial pressure (SAP) to <100 mm Hg. A report led in the UK in 1999 found that most expert obstetric anesthetists utilize a hypotension limit of either 100 or 90 mm Hg of SAP (Šklebar et al., 2019).

General anesthesia GA is either inhaled or injected, causing a state of unconsciousness carefully controlled. It is clinically useful due to its ability to induct rapidly, therefore useful in emergency situations. GA drugs can cross the placenta affecting the fetus. Furthermore, it was commonly believed that it could cause birth asphyxia. GA-induced hypotension was noted as 28% in participants in one study, with systolic and diastolic BP not notably contrasting with the SA group; however, it was more hemodynamically stable and had a minor impact on Apgar score along with umbilical cord blood gas. ICU admissions can happen due to hypotension in GA but less than SA (Alnour et al., 2015; Chen et al., 2019).

Regional anesthesia SA is given for a local anesthetic effect lasting for 2-3 hours; it is widely used. However, rejection by patients for this method is due to anxiety, tension, fear of visualizing the operating room environment, and the thought of being paralyzed. SA-induced hypotension was a research subject for more than 50 years (Alnour et al., 2015; Chen et al., 2019; Šklebar et al., 2019). The decrease in systemic vascular resistance (SVR), which is caused by loss of sympathetic tone in SA reduces CO and SVR. This effect will be compounded by fall in BP due to supine hypotension syndrome (Mavridou et al., 2013). The hypotension rate in SA significantly fluctuates between 7.4% and 74.1%, and in another study, 64% - 100% (Nikooseresht et al., 2016; Šklebar et al., 2019). Hypotension was noted as 48% of participants having CS under SA in a study in Libya (Alnour et al., 2015). Interestingly, it was reported by one of the studies that SA increased CO by 13%, with no significant changes observed in total peripheral resistance (TPR) or mean arterial pressure (MAP) (Ram et al., 2017). Hypotension was also seen in participants undergoing CS with techniques where both SA and EA were used together. (Chen et al., 2019). Prolonged SA-induced hypotension accompanied by decreased SAP can inadequately affect fetal circulation leading to fetal acidosis and hypoxia (Alnour et al., 2015; Šklebar et al., 2019).

There are no studies done to compare GA and RA specifically in terms of the hemodynamic perspective alone (Alnour et al., 2015; Šklebar et al., 2019). Therefore, the present study aimed to find a superior anesthetic technique from a hemodynamic standpoint and proposed a better technique for managing hemodynamic instabilities of pregnant patients undergoing CS.

Aim of this study To examine and find a better technique of anesthesia for the cesarean section from a hemodynamic perspective.

Specific objectives

* To study adverse hemodynamic effects associated with general versus regional anesthetic techniques for cesarean section.
* To propose a superior anesthetic technique from the hemodynamic perspective for cesarean section.

Methodology Setting and design A five-year retrospective cohort study on patients who underwent CS from 1st January 2015 to 31st December 2019 at Sultan Qaboos University Hospital (SQUH) in the Department of Anesthesia and Intensive care, after obtaining ethical approval from the Medical Research committee at SQUH in July 2020 (MREC #2178). The "TrakCare" hospital information system was used to acquire patients' demographic data.

Patients The inclusion criteria of this study were all the patients that underwent CS in SQUH during the study period, and the exclusion criteria were missing data. The sample size of this study included all the patients who underwent CS in this study period, as there were no prior similar studies to calculate the sample size from. A total of 2500 patients were included and coded for identity. This study was not based on any previous studies. Therefore, the population was regarded as all of the patients included in the study period.

Data collection The data was obtained from the hospital information system "TrakCare." Data like age, the urgency of surgery, and the type of anesthesia were all recorded before each surgery, along with the ASA physical status classification system grade. Intraoperative data included heart rate (HR) measured as beats per minute (bpm) and blood pressure (BP) measured as (mm Hg) were obtained from the anesthesia records in the attached Electronic Patient Record (EPR) documents. Blood loss measured in liters (L) and APGAR scores of newborns were also obtained from the surgery notes and clinical notes along with the use of vasopressor intraoperatively. Postoperative anesthesia-related complications were recorded along with the postoperative length of stay (Days) and the mortality of the mother and the baby.

Data analysis Data was collected, and the patient's identity was coded. Individual data coding was done and analyzed using Statistical Package for the Social sciences (SPSS) software (version23). Descriptive statistics were used to present the data. The Chi-Square test was used to determine the association between different variables under investigation with a p-value of <0.05 considered to be statistically significant. Continuous variables were suitably analyzed using means+/- SD. Missing data was ignored if the percentage of the missing data was less than 10%. The graphical representation tools of SPSS software such as bar charts, pie charts, and cross-tabulation were used to describe the analyzed data and present the categorized and uncategorized variables.

ELIGIBILITY:
Inclusion Criteria:

* All the patients that underwent CS in SQUH during the study period (Jan'2015 - Dec'2019)

Exclusion Criteria:

* Patients with missing data

Ages: 17 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All the patients who underwent Cesarean section under either type of Anesthesia, electively or in an emergency situation, with different indications, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | 2-3 hours
  Systolic Blood pressure less than 90 mm hg

SECONDARY OUTCOMES:
Intraoperative blood loss | 2-3 hours
  Effect of type of Anesthesia or it's sequelae on Blood loss during Cesarean section
Impact on APGAR Score | 2-3 hours
  Effect of type of anesthsia or it's sequelae on foetal APGAR score

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD, EDIC, Study Director — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: when summary data are published
Access Criteria: Data might be accessible for any meta-analysis related to the study subject.

REFERENCES:
- See also: Alnour, T. M., et al (2015) Comparison between the Side Effects of Spinal and General Anesthesia during Caesarean Section in Tripoli-Libya. https://doi.org/10.4172/2155-6148.1000560 — https://www.longdom.org/special-issues/obstetric-anesthesia-1475.html
- See also: Aregawi, A., et al. (2018) Comparing the Effect of Spinal and General Anaesthesia for Pre-Eclamptic Mothers Who Underwent Caesarean Delivery in A Tertiary, Addis Ababa, Ethiopia, Ethiopian journal of health sciences. NLM — https://pubmed.ncbi.nlm.nih.gov/30607057/
- See also: Chen, Y., et al. (2019) Comparison of effects of general anesthesia and combined spinal/epidural anesthesia for cesarean delivery on umbilical cord blood gas values: A double-blind, randomized, controlled study, Medical Science Mo. — https://pubmed.ncbi.nlm.nih.gov/31308355/
- See also: Kinzhalova, S.; Makarov, R.; Davidova, N. (2013) Comparison of general and spinal anaesthesia on haemodynamic parameters in severe preeclamptic pregnancy undergoing caesarean section, European Journal of Anaesthesiology. — https://pubmed.ncbi.nlm.nih.gov/25306680/
- See also: Ko, S. (2012) Does choice of anesthetics affect intraoperative blood loss?, Korean Journal of Anesthesiology. Korean Society of Anesthesiologists, 295-296. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3483485/
- See also: tade, A., et al. (2018) Measurements of Inferior Vena Cava Diameter for Prediction of Hypotension and Bradycardia during Spinal Anesthesia in Spontaneously Breathing Patients during Elective Knee Joint Replacement Surgery — https://pubmed.ncbi.nlm.nih.gov/30344280/
- See also: Mavridou, I., Stewart, A. and Fernando, R. (2013) OBSTETRICAL ANESTHESIA (LR LEFFERT, SECTION EDITOR) Maternal Hypotension During Spinal Anesthesia for Cesarean Delivery, Current Anesthesiology Reports 2013 3:4. Springer, 3(4): 282-291. — https://link.springer.com/article/10.1007/s40140-013-0036-3
- See also: Nikooseresht, M., Seif Rabiei, M. A., Hajian, P., Dastaran, R. and Alipour, N. (2016) Comparing the hemodynamic effects of spinal anesthesia in preeclamptic and healthy parturients during cesarean section, Anesthesiology and Pain Medicine. — https://pubmed.ncbi.nlm.nih.gov/27642568/
- See also: Ram, M., et al. (2017) Cardiac hemodynamics before, during and after elective cesarean section under spinal anesthesia in low-risk women, Journal of Perinatology. — https://www.nature.com/articles/jp201753
- See also: Saha, L. and Chowdhury, S. B. (2011) Study on primary cesarean section., Mymensingh medical journal : MMJ. Bangladesh, 20(2): 292-297. — https://pubmed.ncbi.nlm.nih.gov/21522103/
- See also: Šklebar, I., Bujas, T. and Habek, D. (2019) Spinal anaesthesia-induced hypotension in obstetrics: Prevention and therapy, Acta Clinica Croatica. Klinicka Bolnica Sestre Milosrdnice, 58(Suppl 1): 90-95. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6813480/
- See also: Stark, A. R., Adamkin, D. H., Batton, D. G., Bell, E. F., Bhutani, V. K., Denson, S. E., … Hawks, D. (2006) The Apgar score, Pediatrics. American Academy of Pediatrics, 1444-1447. — https://pubmed.ncbi.nlm.nih.gov/16585348/